CLINICAL TRIAL: NCT01474681
Title: A First-in-human, Single-arm, Single-center, Open-label, Proof-of-concept Study to Evaluate the Safety and Tolerability of Infusing HSC835 (LFU835-expanded Umbilical Cord Blood Hematopoietic Stem Cells) in Patients With Hematological Malignancies
Brief Title: Safety and Tolerability of HSC835 in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHSC835X2201
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2019-03

CONDITIONS: Acute Myelocytic Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome; Chronic Lymphocytic Leukemia; Marginal Zone Lymphoma; Follicular Lymphomas; Large-cell Lymphoma; Lymphoblastic Lymphoma; Burkitt's Lymphoma; High Grade Lymphomas; Mantle-cell Lymphoma; Lymphoplasmacytic Lymphoma
Keywords: hematologic malignancies; leukemia; lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Hematologic Neoplasms; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HSC835 (Experimental): HSC835 infusion
  Interventions: Biological: HSC835

INTERVENTIONS:
Biological: HSC835

SUMMARY:
This study evaluated the safety and tolerability of using HSC835 in patients with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis that qualifies them for a DUCBT
* Absence of recent active mold infection
* Adequate organ function
* Availability of eligible donor material

Exclusion Criteria:

* Pregnancy or breastfeeding women and women of child-bearing potential unless two acceptable forms of contraception are being used
* Human immunodeficiency virus (HIV) infection
* Active infection
* Extensive prior chemotherapy
* Prior myeloablative allotransplantation or autologous transplant.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2016-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Minneapolis, Minnesota, United States

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single arm study of HSC835 broken down into 4 subgroups for analyses and 6 subgroups for safety.
Groups:
- SUCBT < 18 Yrs: Single umbilical cord blood transplant(SUCBT) less than 18 yrs
- SUCBT >= 18 Yrs: Single umbilical cord blood transplant (SUCBT) greater than or equal to 18 yrs
- DUCBT < 18 Yrs: Double umbilical cord blood transplant (DUCBT) less than 18 yrs
- DUCBT >= 18 Yrs: Double umbilical cord blood transplant (DUCBT) greater than or equal to 18 yrs
Period: Overall Study
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Started | 1 | 8 | 3 | 15
Completed | 1 | 5 | 1 | 9
Not Completed | 0 | 3 | 2 | 6
Not completed — Death | 0 | 3 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- SUCBT: Single umbilical cord blood transplant (SUCBT) This is the combination of the SUCBT<18 yrs and SUCBT >= 18 yrs
- DUCBT: Double umbilical cord blood transplant (DUCBT) This is the combination of the DUCBT<18 yrs and DUCBT >= 18 yrs
- Total: Total of all reporting groups
Arm/Group | SUCBT | DUCBT | Total
Number analyzed (Participants) | 9 | 18 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (17.18) | 31.3 (13.75) | 32.0 (14.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of HSC835 for Clinical Use Were Measured by Infusional Toxicity (Within First 48 Hours After Transplant) and Absence of Graft Failure After 32 Days in Excess of That Currently Observed With UCBT.
Description: The safety and tolerability of HSC835 for clinical use were measured by infusional toxicity and absence of graft failure in excess of that currently observed with UCBT. Infusional toxicity - AE from transplant until first 48 hours. Administration of the HSC835 expanded CD34-positive cell product, infused over a period of approximately 15 minutes may theoretically cause adverse reactions based on hemodynamic effects, the release of factors like cytokines through administration into the systemic circulation, or acute hypersensitivity, among others.
Time Frame: 32 days
Population: Safety Analysis Set (SAS) comprising all patients who were transplanted is used for analysis of all demographic, safety and engraftment outputs.
Measure: Number; unit: participants
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 1 | 8 | 3 | 15
participants
  Infusional Toxicity 48 hrs after transplant | 0 | 0 | 0 | 1
  Absence of graft failure after 32 days | 0 | 0 | 0 | 0

2. Secondary Outcome: Incidence of Neutrophil Recovery Within 42 Days
Description: Neutrophil recovery (engraftment) is defined as the first of three consecutive days with ANC > 0.5 x 109/L which occurred for all patients before 42 days post transplant.
Time Frame: 42 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 1 | 8 | 3 | 15
participants | 1 | 8 | 3 | 15

3. Secondary Outcome: Incidence of Platelet Recovery Within Six Months
Description: Incidence of platelet recovery within six months. Number of participants recovering platelet to ≥50,000 × 109/L for at least one week without transfusion in the prior 7 days to the first measurement.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 1 | 8 | 3 | 15
participants | 1 | 6 | 2 | 11

4. Secondary Outcome: Frequency of Expanded Unit Predominance at Day 100 (DUCBT Recipients Only)
Description: Frequency of expanded unit predominance at day 100 (DUCBT recipients only) unit predominance was assessed by differences in microsatellite patterns between the recipient, HSC835 and the unmanipulated cord blood unit. Evaluation of sorted CD15-positive/CD33-positive myeloid and CD3-positive T cells in the peripheral blood, revealed three patterns: predominance of HSC835, Mixed dominance an unique chimerism pattern was observed with the CD15/CD33 population predominantly derived from HSC835 and the CD3 population almost exclusively derived from the unmanipulated unit, and predominance of the unmanipulated unit
Time Frame: Day 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 3 | 15
participants
  Predominance of HSC835 | 0 | 6
  Mixed dominance | 3 | 3
  Predominance of the unmaninpulated unit | 0 | 6

5. Secondary Outcome: Incidence of Transplant Related Mortality (TRM) Within 100 Days and One Year
Description: Number of participants with incidence of transplant related mortality (TRM) within 100 days and one year
Time Frame: Day 100 and Month 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 1 | 8 | 3 | 15
participants
  Day 100 | 0 | 1 | 1 | 3
  Month 12 | 0 | 1 | 1 | 6

6. Secondary Outcome: Incidence of Acute Graft Versus Host Disease (aGVHD) Within 100 Days and Chronic Graft Versus Host Disease (cGVHD) Within 1 Year
Description: Number of participants with incidence of Acute Graft Versus Host Disease (aGVHD) within 100 days and Chronic Graft Versus Host Disease (cGVHD) within 1 year
Time Frame: Day 100 and Monnth 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 1 | 8 | 3 | 15
participants
  aGVHD-Day 100 | 0 | 5 | 3 | 8
  cGVHD-Month12 | 0 | 1 | 0 | 2

7. Secondary Outcome: Incidence of Relapse Within One Year
Description: Number of participants with Incidence of relapse within one year
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 1 | 8 | 3 | 15
participants | 0 | 2 | 1 | 0

8. Secondary Outcome: Overall Survival (OS) Within One Year
Description: Number of participants with Overall survival (OS) within one year
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 1 | 8 | 3 | 15
participants | 1 | 5 | 1 | 9

9. Secondary Outcome: Disease Free Survival (DFS) Within One Year
Description: Number of participants with Disease Free Survival (DFS) within one year. Patients are considered to have achieved DFS or relapse-free survival if they had not experienced either relapse or death (of any cause)
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs
Number analyzed (Participants) | 1 | 8 | 3 | 15
participants | 1 | 5 | 1 | 9

ADVERSE EVENTS:
Arm/Group | SUCBT < 18 Yrs | SUCBT >= 18 Yrs | DUCBT < 18 Yrs | DUCBT >= 18 Yrs | SUCBT | DUCBT
Serious Adverse Events (participants affected / at risk) | 1/1 | 7/8 | 3/3 | 14/15 | 8/9 | 17/18
Other Adverse Events (participants affected / at risk) | 1/1 | 8/8 | 3/3 | 15/15 | 9/9 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUCBT < 18 Yrs (N=1) | SUCBT >= 18 Yrs (N=8) | DUCBT < 18 Yrs (N=3) | DUCBT >= 18 Yrs (N=15) | SUCBT (N=9) | DUCBT (N=18)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute graft versus host disease (Immune system disorders) | 0 | 5 | 2 | 8 | 5 | 10
Acute graft versus host disease in skin (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chronic graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 2 | 1 | 2
Engraftment syndrome (Immune system disorders) | 0 | 0 | 0 | 3 | 0 | 3
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
BK virus infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Candida pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Cerebral aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Meningitis enterococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Meningitis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 2 | 1 | 3
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 3
Pneumonia fungal (Infections and infestations) | 0 | 2 | 0 | 2 | 2 | 2
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 2 | 0 | 0 | 2 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Viral myocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 2 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 5 | 0 | 5
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 4 | 2 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Venoocclusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SUCBT < 18 Yrs (N=1) | SUCBT >= 18 Yrs (N=8) | DUCBT < 18 Yrs (N=3) | DUCBT >= 18 Yrs (N=15) | SUCBT (N=9) | DUCBT (N=18)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 12 | 5 | 14
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 1 | 2
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 3 | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 5 | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 3 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 7 | 1 | 10 | 8 | 11
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 0 | 5
Chills (General disorders) | 0 | 1 | 0 | 6 | 1 | 6
Face oedema (General disorders) | 0 | 1 | 1 | 1 | 1 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
BK virus infection (Infections and infestations) | 0 | 3 | 1 | 4 | 3 | 5
Bacillus bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1 | 2 | 1 | 3
Corynebacterium bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 1 | 4 | 0 | 5
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Granulicatella infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Moraxella infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Osteomyelitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 4 | 2 | 6 | 4 | 8
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 3 | 10 | 5 | 13
Fluid overload (Metabolism and nutrition disorders) | 1 | 4 | 1 | 6 | 5 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 4 | 1 | 7 | 4 | 8
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 2 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 6 | 2 | 6
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5 | 1 | 5
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 6 | 1 | 10 | 6 | 11
Hypotension (Vascular disorders) | 0 | 2 | 2 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.